CLINICAL TRIAL: NCT00720278
Title: Randomized, Double-Blind, Placebo-Controlled Trial of the Safety and Efficacy of MP03-36 and MP03-33 Compared to Placebo in Patients With Seasonal Allergic Rhinitis
Brief Title: A Study to Evaluate the Safety and Efficacy of Two Nasal Sprays to Treat Seasonal Allergies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Responsible Party: Harry Sacks, MD Vice President, Medical and Scientific Affairs, Med Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP438
Record Dates: First submitted 2008-07-21; First posted 2008-07-22 (Estimated); Results first posted 2009-10-27 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — azelastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo Nasal Spray (Placebo Comparator): Placebo nasal spray
  Interventions: Drug: Placebo
- Astepro 0.1% (Experimental): 0.1% azelastine hydrochloride nasal spray
  Interventions: Drug: 0.1% azelastine hydrochloride 1096 mcg daily
- Astepro 0.15% (Experimental): 0.15% azelastine hydrochloride nasal spray
  Interventions: Drug: 0.15% azelastine hydrochloride 1644 mcg daily

INTERVENTIONS:
Drug: 0.15% azelastine hydrochloride 1644 mcg daily — 0.15% azelastine hydrochloride 1644 mcg daily
  Other Names: Astepro 0.15%
  Arms: Astepro 0.15%
Drug: 0.1% azelastine hydrochloride 1096 mcg daily — 0.1% azelastine hydrochloride 1096 mcg daily
  Other Names: Astepro 0.1%
  Arms: Astepro 0.1%
Drug: Placebo — 0 mcg Placebo daily
  Arms: Placebo Nasal Spray

SUMMARY:
The purpose of this study was to determine if two allergy medications are more effective than placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 12 years of age and older
2. Provide written informed consent/pediatric assent. If the patient is a minor, a parent or legal guardian must give written informed consent
3. Screening Visit: Have a 12-hour reflective TNSS of at least 8 out of a possible 12 and a congestion score of 2 or 3 on Day -7
4. Randomization Visit: Have a 12-hour reflective TNSS (AM or PM) of at least 8 on 3 separate symptom assessments (one of which was within 2 days of Day 1, and can include the morning of Day 1) during the Lead-in Period. In addition, an AM or PM 12-hour reflective nasal congestion score of 2 or 3 must have been recorded on 3 separate symptom assessments (one of which was within 2 days of Day 1, and can include the morning of Day 1)
5. Randomization Visit: An instantaneous TNSS of ≥ 8 before beginning the onset of action assessment on Day 1
6. Must have taken at least 10 doses of study medication during the lead-in period
7. Willing and able to comply with the study requirements
8. At least a 2-year history of SAR
9. The presence of IgE-mediated hypersensitivity to ragweed antigen or other local fall allergens, confirmed by a positive response to either skin prick within the last year. A positive response is defined as a wheal diameter of at least 3 mm larger than the negative control for the skin prick test.
10. General good health and free of any disease or concomitant treatment that could interfere with the interpretation of the study results as determined by the investigator or the sponsor's medical officer. When in doubt, the investigator should confer with the sponsor's medical monitor or designee to determine eligibility for the study.
11. Patients receiving immunotherapy injections (antigen desensitization) must be on a stable maintenance regimen for at least 30 days before the first study visit (adjustments to regimen following a brief period of missed injections does not preclude participation). Patients currently receiving sublingual immunotherapy are excluded. A 6-month washout period is required following the last dose of sublingual immunotherapy.

Exclusion Criteria:

1. On Focused Nasal Examination, the presence of any nasal mucosal erosion, nasal ulceration, or nasal septal perforation at either the screening visit or randomization visit will disqualify the patient from the study.
2. Other nasal disease(s) likely such as sinusitis, rhinitis medicamentosa, clinically significant polyposis, or nasal structural abnormalities.
3. Nasal surgery or sinus surgery within the previous year.
4. Chronic sinusitis - more than 3 episodes per year
5. Planned travel outside of the study area during the study period
6. The use of any investigational drug within 30 days prior to Day -7. No investigational products are permitted for use during the conduct of this study
7. Presence of any hypersensitivity to drugs similar to azelastine and to either sorbitol or sucralose (Splenda® brand sweetener)
8. Women who are pregnant or nursing
9. Women of childbearing potential who are not abstinent or not practicing a medically acceptable method of contraception
10. Respiratory Tract Infections within 14 days prior to Day -7
11. Respiratory Tract Infections requiring oral antibiotic within 14 days of Day -7
12. Asthma (with the exception of mild, intermittent asthma). Patients with mild, intermittent asthma who only require short-acting inhaled bronchodilators are eligible for enrollment.
13. Significant pulmonary disease including COPD
14. Clinically significant arrhythmia or with symptomatic cardiac conditions
15. A known history of alcohol or drug abuse
16. Existence of any surgical or medical condition or physical or laboratory findings, which in the opinion of the investigator or sponsor's medical monitor, might significantly alter the absorption, distribution, metabolism, or excretion of study drug or that might significantly affect the patient's ability to complete this trial.
17. Clinically relevant abnormal physical findings within 1 week of randomization which, in the opinion of the investigator, would interfere with the objectives of the study or that may preclude compliance with the study procedures
18. Participation in MedPointe Protocols MP433, MP434, MP435, or MP436.
19. Employees of the research center or private practice and their family members are excluded
20. Patients who received prohibited medications within specified timepoints in the protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2007-08; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Center of Research Excellence, LLC, Oxford, Alabama
  - Clinical Research Center, Encinitas, California
  - Allergy Research Foundation, Los Angeles, California
  - Southern California Research, Mission Viejo, California
  - Allergy Associates Medical Group Inc, San Diego, California
  - Storms Clinical Research Institute, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Centers, Denver, Colorado
  - ENTA Allergy, Head and Neck Associates, Decatur, Illinois
  - Sneeze, Wheeze and Itch Associates, Normal, Illinois
  - Family Allergy and Asthma Reserach, Louisville, Kentucky
  - Northeast Medical Research Associates, North Dartmouth, Massachusetts
  - Clinical Research Institute, Plymouth, Minnesota
  - Allergy, Asthma and Immunology Associates, Lincoln, Nebraska
  - Atlantic Research Center, Ocean City, New Jersey
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Research Asthma, Sinus and Allergy Centers, Warren Township, New Jersey
  - AAIR Research Center, Rochester, New York
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Allergy, Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - Allergy and Consultants of NJ/PA, Collegeville, Pennsylvania
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - National Allergy, Asthma and Urticaria of Charleston, Charleston, South Carolina
  - East Tennesse Center for Clinical Research, Knoxville, Tennessee
  - Allergy and Asthma Associates, Austin, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Biogenics Research Institute, San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Allergy and Asthma Care, Waco, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First observation: 14 Aug 2007 Last observation: 19 Nov 2007
Pre-assignment Details: Subjects participated in a 7 day screening period to Identify appropriate subjects based on symptom scores.
Groups:
- Placebo: Placebo Nasal Spray taken 2 sprays per nostril twice a day for 14 days
- Astepro 0.1%: 0.1% azelastine hydrochloride Nasal Spray taken 2 sprays per nostril twice a day for 14 days
- Astepro 0.15%: 0.15% azelastine hydrochloride Nasal Spray taken 2 sprays per nostril twice a day for 14 days
Period: Overall Study
Arm/Group | Placebo | Astepro 0.1% | Astepro 0.15%
Started | 178 (1 subject was randomized in error) | 170 (1 subject was randomized in error) | 178 (1 subject was randomized in error)
Completed | 171 | 166 | 172
Not Completed | 7 | 4 | 6
Not completed — Adverse Event | 5 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Non-compliance | 1 | 0 | 0
Not completed — eligibility criteria violation | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Astepro 0.1% | Astepro 0.15% | Total
Number analyzed (Participants) | 177 | 169 | 177 | 523
Age, Categorical [Count of Participants; unit: Participants] — Number of participants based on ITT population
  Participants
    <=18 years | 24 | 16 | 16 | 56
    Between 18 and 65 years | 148 | 151 | 156 | 455
    >=65 years | 5 | 2 | 5 | 12
Age Continuous [Mean (Standard Deviation); unit: years] — Number of participants based on ITT population
  years | 36.9 (14.27) | 35.4 (13.74) | 37.7 (14.64) | 36.7 (14.23)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of participants based on ITT population
  Participants
    Female | 116 | 111 | 107 | 334
    Male | 61 | 58 | 70 | 189
Region of Enrollment [Number; unit: participants] — Number of participants based on ITT population
  participants
    United States | 177 | 169 | 177 | 523

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 12-hour Reflective Total Nasal Symptom Score(rTNSS)for the Entire 14-day Study Period Compared to Placebo
Description: rTNSS consisting of runny nose, itchy nose, nasal congestion, and sneezing was assessed twice daily. Each symptom is rated on a scale from 0-3: 0=none, 1=mild, 2=moderate, and 3=severe. (maximum 12 points per assessment.) Total possible score is 24 per day.
  Least square means was controlled for study day as the within-patient effect, treatment group and site as the between-patient effects, treatment by-study day interaction, and baseline as a covariate.
Time Frame: baseline and 14 days
Measure: Least Squares Mean (Standard Deviation); unit: total nasal symptom score
Arm/Group | Placebo | Astepro 0.1% | Astepro 0.15%
Number analyzed (Participants) | 171 | 166 | 172
total nasal symptom score
  Baseline symptom score | 17.86 (3.301) | 18.29 (3.23) | 17.83 (3.284)
  Overall change from baseline | -2.36 (4.155) | -4.42 (4.696) | -5.36 (5.077)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.1%; Change in baseline to Day 14; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -2.06, 95% CI [-2.98 to -1.14], Standard Deviation 0.470
Statistical Analysis 2: Comparison: Placebo vs Astepro 0.15%; Change in baseline to Day 14; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -3.00, 95% CI [-3.91 to -2.09], Standard Deviation 0.465

2. Secondary Outcome: Change From Baseline in Instantaneous Total Nasal Symptom Score for the Entire 14-day Study Period Compared to Placebo
Description: instantaneous (subjects rate how they feel "right now") total nasal symptom score consisting of runny nose, itchy nose, nasal congestion, and sneezing was assessed twice daily. Each symptom is rated on a scale from 0-3: 0=none, 1=mild, 2=moderate, and 3=severe. Total possible score is 24 per day.
  Least square means was controlled for study day as the within-patient effect, treatment group and site as the between-patient effects, treatment by-study day interaction, and basline as a covariate.
Time Frame: baseline and 14 Days
Measure: Least Squares Mean (Standard Deviation); unit: total nasal symptom score
Arm/Group | Placebo | Astepro 0.1% | Astepro 0.15%
Number analyzed (Participants) | 171 | 166 | 172
total nasal symptom score
  Baseline symptom score | 16.56 (3.962) | 17.22 (3.836) | 16.43 (3.998)
  Overall change from baseline | -1.96 (4.313) | -3.74 (4.796) | -4.63 (5.261)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.1%; Change in baseline to Day 14; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -1.78, 95% CI [-2.72 to -0.84], Standard Deviation 0.479
Statistical Analysis 2: Comparison: Placebo vs Astepro 0.15%; Change in baseline to Day 14; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -2.668, 95% CI [-3.60 to -1.74], Standard Deviation 0.4735

3. Secondary Outcome: Change From Baseline in the 12-hour Reflective Secondary Symptom Complex Score for the Entire 14-day Study Period Compared to Placebo
Description: Reflective secondary symptom scores (SSCS) (post-nasal drip, itchy eyes, cough and headache) were assessed twice daily. Each symptom is rated on a scale from 0-3: 0=none, 1=mild, 2=moderate, and 3=severe. Total possible SSCS score is 24 per day.
  Least square means was controlled for study day as the within-patient effect, treatment group and site as the between-patient effects, treatment by-study day interaction, and basline as a covariate.
Time Frame: baseline and 14 days
Measure: Least Squares Mean (Standard Deviation); unit: Reflective secondary symptom score
Arm/Group | Placebo | Astepro 0.1% | Astepro 0.15%
Number analyzed (Participants) | 171 | 166 | 172
Reflective secondary symptom score
  Baseline SSCS | 14.27 (4.503) | 14.59 (4.818) | 13.59 (5.087)
  Change in baseline to Day 14 | -1.72 (3.823) | -3.09 (4.337) | -4.15 (4.600)
Statistical Analysis 1: Comparison: Placebo vs Astepro 0.1%; Change in baseline to Day 14; Test type: Superiority or Other; p = 0.001, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -1.376, 95% CI [-2.20 to -0.56], Standard Deviation 0.418
Statistical Analysis 2: Comparison: Placebo vs Astepro 0.15%; Change in baseline to Day 14; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA is being used due to a covariate being included in the model. The covariate is baseline TNSS score; Mean Difference (Final Values) = -2.432, 95% CI [-3.24 to -1.62], Standard Deviation 0.4145

4. Secondary Outcome: Change From Baseline to Day 14 in the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Compared to Placebo in Patients 18 Years of Age and Older
Description: A 28-item RQLQ was completed on Day 1 and Day 14 or Early temination. The RQLQ consists of 7 domains rated on a 7 point scale with 0 being not troubled by the allergy symptoms, and 6 being extremely troubled/all of the time.
  Domain score will be calculated from the mean score of all items in the domain. Overall score will be calculated from the mean score of all items.
Time Frame: baseline and 14 days
Measure: Least Squares Mean (Standard Deviation); unit: 28 item/7 domain RQLQ on 0-6 scale
Arm/Group | Placebo | Astepro 0.1% | Astepro 0.15%
Number analyzed (Participants) | 171 | 166 | 172
28 item/7 domain RQLQ on 0-6 scale
  Baseline: Overall | 3.87 (0.991) | 3.73 (0.998) | 3.75 (1.012)
  Change from Baseline:Overall | -0.94 (1.112) | -1.12 (1.246) | -1.48 (1.328)

5. Secondary Outcome: Change From Baseline on Direct Visual Nasal Exams
Description: Examination of head and neck (scale: None, Mild, Moderate, Severe) for Epistaxis, Mucosal Edema, Nasal Discharge, Mucosal erythema, Mucosal Bleeding, and Crusting of mucosa.
  Nasal irratation was rated: 0 = None, Grade 1A = focal irritation, Grade 1B = superficial mucosal erosion, Grade 2 = moderate mucosal erosion, Grade 3 = ulceration, Grade 4 = septal perforation
Time Frame: 14 days
Measure: Number; unit: Participants
Arm/Group | Placebo | Astepro 0.1% | Astepro 0.15%
Number analyzed (Participants) | 171 | 166 | 172
Participants
  Epistaxis: screening - total | 178 | 170 | 178
  Epistaxis: screening - None | 176 | 169 | 176
  Epistaxis: screening - Mild | 2 | 1 | 2
  Epistaxis: screening - Moderate | 0 | 0 | 0
  Epistaxis: screening - Severe | 0 | 0 | 0
  Epistaxis: Day 14/ET - total | 178 | 169 | 175
  Epistaxis: Day 14/ET - None | 174 | 168 | 166
  Epistaxis: Day 14/ET - Mild | 4 | 1 | 9
  Epistaxis: Day 14/ET - Moderate | 0 | 0 | 0
  Epistaxis: Day 14/ET - Severe | 0 | 0 | 0
  Nasal Irritation: screening - total | 178 | 0 | 0
  Nasal Irritation: screening - None | 169 | 170 | 178
  Nasal Irritation: screening - Grade 1A | 0 | 166 | 169
  Nasal Irritation: screening - Grade 1B | 0 | 4 | 9
  Nasal Irritation: screening - Grade 2 | 0 | 0 | 0
  Nasal Irritation: screening - Grade 3 | 0 | 0 | 0
  Nasal Irritation: screening - Grade 4 | 0 | 0 | 0
  Nasal Irritation: Day 14/ET - Total | 178 | 169 | 175
  Nasal Irritation: Day 14/ET - None | 168 | 161 | 165
  Nasal Irritation: Day 14/ET- Grade 1A | 8 | 8 | 7
  Nasal Irritation: Day 14/ET- Grade 1B | 2 | 0 | 3
  Nasal Irritation: Day 14/ET- Grade 2 | 0 | 0 | 0
  Nasal Irritation: Day 14/ET- Grade 3 | 0 | 0 | 0
  Nasal Irritation: Day 14/ET- Grade 4 | 0 | 0 | 0
  Mucosal Edema: screening - Total | 178 | 170 | 178
  Mucosal Edema: screening - None | 3 | 3 | 3
  Mucosal Edema: screening - Mild | 40 | 30 | 28
  Mucosal Edema: screening - Moderate | 108 | 106 | 114
  Mucosal Edema: screening - Severe | 27 | 31 | 33
  Mucosal Edema: Day 14/ET - total | 178 | 169 | 175
  Mucosal Edema: Day 14/ET - None | 14 | 12 | 15
  Mucosal Edema: Day 14/ET - Mild | 50 | 60 | 59
  Mucosal Edema: Day 14/ET - Moderate | 88 | 77 | 81
  Mucosal Edema: Day 14/ET - Severe | 26 | 20 | 20
  Nasal Discharge: screening - Total | 178 | 170 | 178
  Nasal Discharge: screening - None | 29 | 26 | 28
  Nasal Discharge: screening - Mild | 72 | 63 | 67
  Nasal Discharge: screening - Moderate | 64 | 67 | 71
  Nasal Discharge: screening - Severe | 13 | 14 | 12
  Nasal Discharge: Day 14/ET - Total | 178 | 169 | 175
  Nasal Discharge: Day 14/ET - None | 26 | 46 | 47
  Nasal Discharge: Day 14/ET- Mild | 85 | 71 | 72
  Nasal Discharge: Day 14/ET - Moderate | 47 | 46 | 45
  Nasal Discharge: Day 14/ET - Severe | 10 | 6 | 11
  Mucosal Erythema: screening - Total | 178 | 170 | 178
  Mucosal Erythema: screening - None | 81 | 74 | 92
  Mucosal Erythema: screening - Mild | 59 | 56 | 45
  Mucosal Erythema: screening - Moderate | 37 | 37 | 39
  Mucosal Erythema: screening - Severe | 1 | 3 | 2
  Mucosal Erythema: Day 14/ET - Toal | 178 | 167 | 175
  Mucosal Erythema: Day 14/ET - None | 101 | 97 | 105
  Mucosal Erythema: Day 14/ET - Mild | 51 | 49 | 42
  Mucosal Erythema: Day 14/ET - Moderate | 25 | 18 | 27
  Mucosal Erythema: Day 14/ET - Severe | 1 | 5 | 1
  Mucosal Bleeding: screening - Toal | 178 | 170 | 178
  Mucosal Bleeding: screening - None | 175 | 167 | 167
  Mucosal Bleeding: screening - Mild | 3 | 3 | 2
  Mucosal Bleeding: screening - Moderate | 0 | 0 | 0
  Mucosal Bleeding: screening - Severe | 0 | 0 | 0
  Mucosal Bleeding: Day 14/ET - Total | 178 | 169 | 175
  Mucosal Bleeding: Day 14/ET - None | 171 | 163 | 163
  Mucosal Bleeding: Day 14/ET - Mild | 7 | 6 | 11
  Mucosal Bleeding: Day 14/ET - Moderate | 0 | 0 | 0
  Mucosal Bleeding: Day 14/ET - Severe | 0 | 0 | 1
  Crusting of Mucosa: screening - Total | 178 | 170 | 178
  Crusting of Mucosa: screening - None | 156 | 142 | 158
  Crusting of Mucosa: screening - Mild | 17 | 20 | 18
  Crusting of Mucosa: screening - Moderate | 4 | 7 | 2
  Crusting of Mucosa: screening - Severe | 1 | 1 | 0
  Crusting of Mucosa: Day 14/ET - Total | 178 | 169 | 175
  Crusting of Mucosa: Day 14/ET - None | 154 | 148 | 155
  Crusting of Mucosa: Day 14/ET - Mild | 19 | 19 | 16
  Crusting of Mucosa: Day 14/ET - Moderate | 4 | 2 | 3
  Crusting of Mucosa: Day 14/ET - Severe | 1 | 0 | 1

ADVERSE EVENTS:
Arm/Group | Placebo | Astepro 0.1% | Astepro 0.15%
Serious Adverse Events (participants affected / at risk) | 2/178 | 0/170 | 0/178
Other Adverse Events (participants affected / at risk) | 5/178 | 21/170 | 19/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=178) | Astepro 0.1% (N=170) | Astepro 0.15% (N=178)
Exposure in utero (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=178) | Astepro 0.1% (N=170) | Astepro 0.15% (N=178)
Dysgesusia (Nervous system disorders) | 2 (2) | 16 (16) | 15 (15)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multicenter studies, joint publication is required to assure that the initial publication is based on all data from all sites and investigators participating in these studies agree not to present data gathered individually or by subgroup centers before the initial publication unless jointly agreed by all other investigators and the sponsor. authorship will be determined by mutual agreement.